CLINICAL TRIAL: NCT03470064
Title: Early Right Ventricular Function After Repair Of Tetralogy Of Fallot , An Evidence Based Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ehab abd-alaal zahran, Assistant lecturer at cardiothoracic surgery department, Assiut University
Other Study IDs: 17200175
Record Dates: First submitted 2018-03-03; First posted 2018-03-19 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RV Dysfunction: All pediatric patients who present to pediatric cardiothoracic unit, Assiut University Hospital and who meet the listed inclusion and exclusion criteria will be eligible for the study. Patients' charts will be retrieved based on their surgical procedures. The charts will be reviewed and eligible patients will be filtered. The needed variables will be entered into our data base for later data analysis

SUMMARY:
This study aims to assessing right ventricular function early after surgical repair of tetralogy of Fallot and identifying the risk factors associated with development of RV dysfunction.

DETAILED DESCRIPTION:
The shape of the RV is dramatically modified by surgical repair of CHD, with infundibular bulging and apical dilation and deformation, leading to a large range of RV shapes(1,2). Moreover, pericardial section and suture during surgery influence RV geometry, as RV is normally more con-strained by the pericardium then the LV because of its thinner wall (3).

Intra cardiac repair(ICR) is the definitive management of TOF. Refinement in surgical techniques, advancements in anaesthetic & critical care has resulted in improving survival following ICR. Post operative mortality following ICR is reported between 1% - 5% (3). Post operative low cardiac output and mortality has been attributed to many factors such as anatomical defects with small main pulmonary artery annulus, severe hypoplasia or absent right or left pulmonary artery, ventriculotomy and right ventricular (RV) outflow patch, myocardial hypoxia during cardiopulmonary bypass, or ARDS (4). Certain patients despite satisfactory ICR exhibit difficult post operative course which is characterized by prolonged ventilation & inotropic support. These patients have been identified to exhibit features of RV dysfunction (low cardiac output, high central venous filling pressure, increased inotropic requirement, and prolonged ventilation). Identification of risk factors to characterise this subset of patients allows for better allocation of hospital resources, improved outcome, and substantially reduced hospital costs. This study will try to identify the risk factors associated with development of RV dysfunction & its course over a period of three months in patients of tetralogy following ICR.

MRI is a gold standard for assessment of right ventricular function (5). However, MRI has restricted availability, is costly, and there are many patients in whom MRI-non compatible devices prohibit its use.

Because of its complex shape, there is no geometrical assumption that can allow quantification of RV volumes and ejection fraction (RVEF) by standard two-dimensional (2D) echocardiography. For this reason, surrogate parameters of RV systolic function are used most frequently to assess RV systolic function, because they are easy to measure, feasible and reproducible. These parameters include:-

* Tricuspid annulus movement:- Measurements of tricuspid annulus movement by M-mode (tricuspid annular plane systolic excursion [TAPSE]) or tissue Doppler imaging (peak systolic velocity [PSV]) are used most frequently to assess RV function; they are highly feasible and reproducible. However, several studies have shown their dependence on loading condition; TAPSE and PSV values are increased in volume overload and decreased in pressure overload (6), independent of RVEF.

-2D global longitudinal peak systolic strain of the RV lateral wall:- Speckle-tracking echocardiography is a new technology that allows quantification of myocardial regional deformation. The main advantage compared with tissue Doppler imaging is its angle independency; it was also thought to be less load dependent, but further studies demonstrated that 2D longitudinal strain values increase in volume overload and decrease in barometric overload (7).

- Isovolumic acceleration time(IVA):- Is a quantitative assessment of RV contractile function that is supposed to be unaffected by RV geometry or loading conditions. In patients with tetralogy of Fallot, studies have shown a good correlation between pulmonary regurgitation severity and IVA (8,9).

-Myocardial performance index :- Myocardial performance index (MPI) is another tissue Doppler-derived parameter of RV systolic function. MPI is calculated using the following formula: MPI =(isovolumic contraction time + isovolumic relaxation time)/ejection time (10).

- Fractional area change:- FAC has been shown to correlate well with RVEF measured by MRI in the general population (10).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients up to 12 years old.
2. Recent echocardiography before the surgery giving detailed data about the components congenital anomalies of tetralogy of Fallot and if there are other associated congenital anomalies.
3. Obtaining written informed consent from parents or guardians of all patients confirming their willing and comply with study requirements
4. Parents or guardians of the Patient are willing to comply with all follow-up visits.

Exclusion Criteria:

1. Patients with tetralogy of Fallot who are indicated to palliative procedures and not for definitive surgical repair as in case of:-

   * Neonates with TOF and pulmonary atresia
   * Children with hypoplastic pulmonary artery
   * Age less than 3 months who have medically unmanageable hypoxic spells
   * Infant weight less than 2.5 kg
   * Abnormal coronary artery anatomy
2. Patients with TOF who are contraindicated to primary repair as in case of:-

   * Multiple VSDs
   * Multiple coexisting intracardiac malformations
   * Small pulmonary arteries
   * Very low birth weight
   * The presence of an anomalous coronary artery
3. Patient inaccessible for follow-up visits required by protocol.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Pediatric patients up to 12 years old.
  2. Recent echocardiography before the surgery giving detailed data about the components congenital anomalies of tetralogy of Fallot and if there are other associated congenital anomalies.
  3. Obtaining written informed consent from parents or guardians of all patients confirming their willing and comply with study requirements
  4. Parents or guardians of the Patient are willing to comply with all follow-up visits
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of RV function early after surgical repair of tetralogy of fallot | within one week postoperative
  the study aim to assess the function of the Right ventricle early after surgical repair of tetralogy of fallot by echocardiography.

SECONDARY OUTCOMES:
Follow up the course of RV function over a period of three months in patients of tetralogy of fallot following surgical repair . | 3 months postoperative
  the study aim to follow up the function of the Right ventricle after surgical repair of tetralogy of fallot by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Zahran, PHD, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
This study aims to assessing right ventricular function early after surgical repair of tetralogy of Fallot and identifying the risk factors associated with development of RV dysfunction.

REFERENCES:
- [Background] Tamborini G, Muratori M, Brusoni D, Celeste F, Maffessanti F, Caiani EG, Alamanni F, Pepi M. Is right ventricular systolic function reduced after cardiac surgery? A two- and three-dimensional echocardiographic study. Eur J Echocardiogr. 2009 Jul;10(5):630-4. doi: 10.1093/ejechocard/jep015. Epub 2009 Feb 27. PMID 19252190
- [Background] Eroglu AG, Sarioglu A, Sarioglu T. Right ventricular diastolic function after repair of tetralogy of Fallot: its relationship to the insertion of a 'transannular' patch. Cardiol Young. 1999 Jul;9(4):384-91. PMID 10476828
- [Background] Higgins CB. Which standard has the gold? J Am Coll Cardiol. 1992 Jun;19(7):1608-9. doi: 10.1016/0735-1097(92)90626-x. No abstract available. PMID 1534338
- [Background] Carminati M, Pluchinotta FR, Piazza L, Micheletti A, Negura D, Chessa M, Butera G, Arcidiacono C, Saracino A, Bussadori C. Echocardiographic assessment after surgical repair of tetralogy of fallot. Front Pediatr. 2015 Feb 2;3:3. doi: 10.3389/fped.2015.00003. eCollection 2015. PMID 25699243
- [Background] Jategaonkar SR, Scholtz W, Butz T, Bogunovic N, Faber L, Horstkotte D. Two-dimensional strain and strain rate imaging of the right ventricle in adult patients before and after percutaneous closure of atrial septal defects. Eur J Echocardiogr. 2009 Jun;10(4):499-502. doi: 10.1093/ejechocard/jen315. Epub 2009 Jan 20. PMID 19155264
- [Background] Frigiola A, Redington AN, Cullen S, Vogel M. Pulmonary regurgitation is an important determinant of right ventricular contractile dysfunction in patients with surgically repaired tetralogy of Fallot. Circulation. 2004 Sep 14;110(11 Suppl 1):II153-7. doi: 10.1161/01.CIR.0000138397.60956.c2. PMID 15364855
- [Background] Eidem BW, O'Leary PW, Tei C, Seward JB. Usefulness of the myocardial performance index for assessing right ventricular function in congenital heart disease. Am J Cardiol. 2000 Sep 15;86(6):654-8. doi: 10.1016/s0002-9149(00)01047-x. PMID 10980218
- [Background] Anavekar NS, Gerson D, Skali H, Kwong RY, Yucel EK, Solomon SD. Two-dimensional assessment of right ventricular function: an echocardiographic-MRI correlative study. Echocardiography. 2007 May;24(5):452-6. doi: 10.1111/j.1540-8175.2007.00424.x. PMID 17456062
- [Background] Wheeler M, Leipsic J, Trinh P, Raju R, Alaamri S, Thompson CR, Moss R, Munt B, Kiess M, Grewal J. Right Ventricular Assessment in Adult Congenital Heart Disease Patients with Right Ventricle-to-Pulmonary Artery Conduits. J Am Soc Echocardiogr. 2015 May;28(5):522-32. doi: 10.1016/j.echo.2014.11.016. Epub 2015 Jan 30. PMID 25648672
- [Background] Leonardi B, Taylor AM, Mansi T, Voigt I, Sermesant M, Pennec X, Ayache N, Boudjemline Y, Pongiglione G. Computational modelling of the right ventricle in repaired tetralogy of Fallot: can it provide insight into patient treatment? Eur Heart J Cardiovasc Imaging. 2013 Apr;14(4):381-6. doi: 10.1093/ehjci/jes239. Epub 2012 Nov 20. PMID 23169758